CLINICAL TRIAL: NCT05134103
Title: A 12-week Randomized Waitlist-Controlled Trial of Mindbeacon Therapist Assisted Internet Delivered CBT for Depression
Brief Title: Mindbeacon Therapist Assisted Internet Delivered CBT for Depression
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor pulled out of study
Sponsor: Ontario Shores Centre for Mental Health Sciences (Other)
Collaborators: Mindbeacon (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 21-004-B
Record Dates: First submitted 2021-10-05; First posted 2021-11-24 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Major Depressive Disorder
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: This is a waitlist-controlled, randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindbeacon TAI-CBT for Depression group (Experimental): Participants randomized to this condition will receive immediate Therapist-Guided Internet-CBT for Depression for 12 weeks.
  Interventions: Behavioral: Mindbeacon Therapist Guided, Internet Cognitive Behavioral Therapy for Depression
- Waitlist Control Group (Other): Participants randomized to this condition will remain on the waitlist for 12 weeks before crossing over and receiving Therapist-Guided Internet-CBT for Depression for 12 weeks.
  Interventions: Other: Waitlist Control Group

INTERVENTIONS:
Behavioral: Mindbeacon Therapist Guided, Internet Cognitive Behavioral Therapy for Depression — The treatment consists of 11 depression modules delivered approximately once per week (at therapists' discretion) over a period of 12 weeks. Additionally, the therapist typically tailors treatment to client's individual needs by including supplementary modules for a variety of issues such as generalized anxiety, panic, social anxiety, post-traumatic stress, insomnia, pain, and relationships etc. Clients can complete the readings, exercises, and worksheets at any convenient time, using their web-enabled smartphone, tablet, or computer. Access to the modules and all messaging is provided through the secure platform. Messaging is "asynchronous" meaning participants can message their therapist as often as they choose and expect a response within 1-2 business days. After 12 weeks of active treatment, they will have unguided access (without therapist support) to the treatment materials that were covered for an additional 40 weeks.
  Other Names: Internet-CBT
  Arms: Mindbeacon TAI-CBT for Depression group
Other: Waitlist Control Group — Participants assigned to this arm will wait for 12 weeks before receiving active treatment condition
  Arms: Waitlist Control Group

SUMMARY:
Utilization of therapist Assisted internet-delivered cognitive behavioural therapy (TAiCBT) for treating depression and anxiety disorders in stepped-care models, such as the UK's Improving Access to Psychological Therapies (IAPT) and the Ontario Structured Psychotherapy Program (SPP), is a potential solution for addressing the treatment gap in mental health. Investigators propose to investigate the effectiveness of Beacon TAiCBT for Depression to demonstrate the potential value of TAiCBT in a stepped care model. Investigators propose to conduct a 12-week pragmatic randomized controlled trial with a 1:1 (iCBT intervention: waiting-list) allocation, for participants referred to the Anxiety and Mood, Prompt Anxiety and Mood, and Trauma Programs at Ontario Shores Centre for Mental Health Sciences and on a waiting-list to receive clinical service.

The primary outcome measures will be the Improving Access to Psychological Therapies (IAPT) definitions of Recovery, Reliable Improvement, and Reliable Recovery which are derived using the PHQ-9 and GAD-7 . The PHQ-9 (Depression), GAD-7 (anxiety) and WSAS (functional impairment) will be used as secondary outcome measures for all participants.

Over the course of the study, 200 participants will be randomized (iCBT, 100; waiting-list, 100). Statistical analyses will include intention-to-treat analyses to test the interaction effects for the primary outcome measures at discharge/12-weeks and 3, and 12 months post-treatment.

It is predicted that participants in the treatment condition will show significantly reduced symptoms of depression related to the waitlist control. It is predicted that this will be maintained through follow up.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Meets Diagnostic Assessment Research Tool (DART) screening criteria for a primary diagnosis of depression and reports being at least moderately depressed according to the PHQ-9
* Sufficient language proficiency to understand the treatment materials written at grade 10 reading level
* Understands what TAiCBT and is open and interested to participating in a study using this treatment modality
* Is able to reliably access the internet, and has basic computer skills to navigate the internet using a web browser
* Willing to participate in a waitlist-control study and be followed for 12 months

Exclusion Criteria:

* Suicidal intent or clinically significant suicidal ideation
* Clinically significant self-harm
* Active psychotic illness
* Currently participating in psychological treatment for depression and/or receiving evidence-based treatment (other than medication) for depression
* Clinically significant alcohol and/or other substance use including prescription and over the counter medication that would likely interfere with treatment
* Current or previous diagnosis of Borderline Personality Disorder
* Does not meet DART criteria for a primary diagnosis of depression
* Change in psychotropic medication within 3 weeks of treatment baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
IAPT Definition of "Recovery" (Change between Baseline and Post-treatment) | GAD-7 and PHQ-9 which are used to compute this outcome measure are administered at baseline (initial screening) and "post-treatment" which is week 12 of treatment)
  The IAPT criteria for 'Recovery' are met when patients move from 'caseness' at the beginning of the intervention (e.g., scoring >9 on the PHQ-9 or >7 on the GAD-7) to 'non-caseness' at the end of treatment (thus scoring below the cut-off)
IAPT Definition of "Recovery" (Change between baseline and 3 month follow-up) | GAD-7 and PHQ-9 which are used to compute this outcome measure are administered at baseline (initial screening) and 3 month follow-up (3 months after "post-treatment" which is week 12 of treatment)
  The IAPT criteria for 'Recovery' are met when patients move from 'caseness' at the beginning of the intervention (e.g., scoring >9 on the PHQ-9 or >7 on the GAD-7) to 'non-caseness' at the end of treatment (thus scoring below the cut-off)
IAPT Definition of "Recovery" (Change between baseline and 12 month follow-up) | GAD-7 and PHQ-9 which are used to compute this outcome measure are administered at baseline (initial screening) and 12 month follow-up (12 months after "post-treatment" which is week 12 of treatment)
  The IAPT criteria for 'Recovery' are met when patients move from 'caseness' at the beginning of the intervention (e.g., scoring >9 on the PHQ-9 or >7 on the GAD-7) to 'non-caseness' at the end of treatment (thus scoring below the cut-off)
IAPT Definition of "Reliable improvement" (Change between Baseline and Post-treatment) | GAD-7 and PHQ-9 which are used to compute this outcome measure are administered at baseline (initial screening) and "post-treatment" which is week 12 of treatment)
  Reliable improvement is defined as when the patient has a 'reliable' decrease in their PHQ-9 / GAD-7 (reduction in PHQ-9 score of 6 or more, and reduction in GAD-7 score of 4 or more) score upon completion of their course of treatment
IAPT Definition of "Reliable improvement" (Change between baseline, and 3 month follow-up) | GAD-7 and PHQ-9 which are used to compute this outcome measure are administered at baseline (initial screening) and 3 month follow-up (3 months after "post-treatment" which is week 12 of treatment)
  Reliable improvement is defined as when the patient has a 'reliable' decrease in their PHQ-9 / GAD-7 (reduction in PHQ-9 score of 6 or more, and reduction in GAD-7 score of 4 or more) score upon completion of their course of treatment
IAPT Definition of "Reliable improvement" (Change between baseline and 12 month follow-up) | GAD-7 and PHQ-9 which are used to compute this outcome measure are administered at baseline (initial screening) and 12 month follow-up (12 months after "post-treatment" which is week 12 of treatment)
  Reliable improvement is defined as when the patient has a 'reliable' decrease in their PHQ-9 / GAD-7 (reduction in PHQ-9 score of 6 or more, and reduction in GAD-7 score of 4 or more) score upon completion of their course of treatment
IAPT definition of "Reliable recovery" (Change between Baseline and Post-treatment) | GAD-7 and PHQ-9 which are used to compute this outcome measure are administered at baseline (initial screening) and post-treatment (week 12 of treatment)
  Reliable recovery is defined as when the patient meets the criteria for both recovery and reliable improvement as defined above. Thus, a patient who moves from caseness to non-caseness, and also shows a 'reliable' (reduction in PHQ-9 score of 6 or more, and reduction in GAD-7 score of 4 or more) decrease in their symptom scores, is said to have a reliable recovery
IAPT definition of "Reliable recovery" (Change between baseline and 3 month follow-up) | GAD-7 and PHQ-9 which are used to compute this outcome measure are administered at baseline (initial screening) and 3 month follow-up (3 months after "post-treatment" which is week 12 of treatment)
  Reliable recovery is defined as when the patient meets the criteria for both recovery and reliable improvement as defined above. Thus, a patient who moves from caseness to non-caseness, and also shows a 'reliable' (reduction in PHQ-9 score of 6 or more, and reduction in GAD-7 score of 4 or more) decrease in their symptom scores, is said to have a reliable recovery
IAPT definition of "Reliable recovery" (Change between baseline and 12 month follow-up) | GAD-7 and PHQ-9 which are used to compute this outcome measure are administered at baseline (initial screening) and 12 month follow-up (12 months after "post-treatment" which is week 12 of treatment)
  Reliable recovery is defined as when the patient meets the criteria for both recovery and reliable improvement as defined above. Thus, a patient who moves from caseness to non-caseness, and also shows a 'reliable' (reduction in PHQ-9 score of 6 or more, and reduction in GAD-7 score of 4 or more) decrease in their symptom scores, is said to have a reliable recovery

SECONDARY OUTCOMES:
Work and Social Adjustment Scale (WSAS) - (Change between Baseline and Post-treatment) | Administered at baseline (initial screening) and post-treatment (week 12 of treatment)
  This is a simple, reliable and valid measure of impaired functioning. It is a 5-item self-report measure that provides an experiential impact of a disorder from the patient's point of view. It looks at how the disorder impairs the patient's ability to function day to day on five dimensions: work, social life, home life, private life and close relationships. This scale ranges from 0-40 with 40 indicating a severe level of functional impairment.
Work and Social Adjustment Scale (WSAS) - (Change between baseline and 3 month follow-up) | Administered at baseline (initial screening) and 3 month follow-up (3 months after "post-treatment" which is week 12 of treatment)
  This is a simple, reliable and valid measure of impaired functioning. It is a 5-item self-report measure that provides an experiential impact of a disorder from the patient's point of view. It looks at how the disorder impairs the patient's ability to function day to day on five dimensions: work, social life, home life, private life and close relationships. This scale ranges from 0-40 with 40 indicating a severe level of functional impairment.
Work and Social Adjustment Scale (WSAS) - (Change between baseline and 12 month follow-up) | Administered at baseline (initial screening) and 12 month follow-up (12 months after "post-treatment" which is week 12 of treatment)
  This is a simple, reliable and valid measure of impaired functioning. It is a 5-item self-report measure that provides an experiential impact of a disorder from the patient's point of view. It looks at how the disorder impairs the patient's ability to function day to day on five dimensions: work, social life, home life, private life and close relationships. This scale ranges from 0-40 with 40 indicating a severe level of functional impairment.
Patient Health Questionnaire 9 (PHQ-9) - (Change between baseline and post-treatment) | Administered at baseline (initial screening) and post-treatment (week 12 of treatment)
  Items on the PHQ-9 reflect symptoms of Major Depressive Disorder, and provides a dimensional measure of symptom severity, self-administered by participants. Scores on this scale range from 0-27 with higher scores indicating more severe depression.
Patient Health Questionnaire 9 (PHQ-9) - (Change between baseline and 3 month follow-up) | Administered at baseline (initial screening) and 3 month follow-up (3 months after "post-treatment" which is week 12 of treatment)
  Items on the PHQ-9 reflect symptoms of Major Depressive Disorder, and provides a dimensional measure of symptom severity, self-administered by participants. Scores on this scale range from 0-27 with higher scores indicating more severe depression.
Patient Health Questionnaire 9 (PHQ-9) - (Change between baseline and 12 month follow-up) | Administered at baseline (initial screening) and 12 month follow-up (12 months after "post-treatment" which is week 12 of treatment)
  Items on the PHQ-9 reflect symptoms of Major Depressive Disorder, and provides a dimensional measure of symptom severity, self-administered by participants. Scores on this scale range from 0-27 with higher scores indicating more severe depression.
Generalized Anxiety Disorder 7 (GAD-7) - (Change between baseline and post-treatment) | Administered at baseline (initial screening) and post-treatment (week 12 of treatment)
  Items on the GAD-7 reflect symptoms of Generalized Anxiety Disorder, and provides a dimensional measure of symptom severity, self-administered by participants. Scores on this scale range from 0-21 with higher scores indicating more severe anxiety.
Generalized Anxiety Disorder 7 (GAD-7) - (Change between baseline and 3 month follow-up) | Administered at baseline (initial screening) and 3 month follow-up (3 months after "post-treatment" which is week 12 of treatment)
  Items on the GAD-7 reflect symptoms of Generalized Anxiety Disorder, and provides a dimensional measure of symptom severity, self-administered by participants. Scores on this scale range from 0-21 with higher scores indicating more severe anxiety.
Generalized Anxiety Disorder 7 (GAD-7) - (Change between baseline and 12 month follow-up) | Administered at baseline (initial screening) and 12 month follow-up (12 months after "post-treatment" which is week 12 of treatment)
  Items on the GAD-7 reflect symptoms of Generalized Anxiety Disorder, and provides a dimensional measure of symptom severity, self-administered by participants. Scores on this scale range from 0-21 with higher scores indicating more severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Phil Klassen, MD, Principal Investigator — Ontario Shores Hospital

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared with other researchers. Anonymized/deidentified aggregate data for the study may be shared.